CLINICAL TRIAL: NCT01569529
Title: Increasing Young Adult Smoker's Demand for Internet-based Cessation Treatment
Brief Title: Young Adult Smoker's Treatment Demand
Status: Completed | Type: Observational
Sponsor: University of Illinois at Chicago (Other)
Collaborators: National Cancer Institute (NCI) (NIH); University of Iowa (Other); Truth Initiative (Other)
Responsible Party: Principal Investigator, Robin Mermelstein, Director, Institute for Health Research and Policy, University of Illinois at Chicago
Other Study IDs: 2008-06778; R01CA134861-01A1 (NIH)
Record Dates: First submitted 2012-03-30; First posted 2012-04-03 (Estimated); Results first posted 2014-05-13 (Estimated); Last update posted 2017-03-30 (Actual); Status verified 2017-02

CONDITIONS: Smoking Cessation
MeSH Terms: conditions — Smoking Cessation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- No ad exposure: Young adults, who enroll in the cessation program, one month prior to presenting the online advertisements (intervention).
- Ad exposure: Young Adults, who register for the cessation program, by clicking through the online advertisements (intervention).
  Interventions: Behavioral: Online advertisement

INTERVENTIONS:
Behavioral: Online advertisement — Internet advertisement with messages tailored for young adult smoker's motivated to quit
  Groups: Ad exposure

SUMMARY:
The purpose of this study is to determine whether tailored online advertisements will drive young adult smoker's (18 to 26 years old), who are motivated to quit, to use Internet-based cessation treatment.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 30 years old
* smoke on some days or everyday
* enrollment in specified online cessation program

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Young adult Internet users
Sampling Method: Non-Probability Sample
Enrollment: 3070 (Actual)
Dates: Start 2012-05; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robin J Mermelstein, PhD, Principal Investigator — University of Illinois at Chicago; Susan J Curry, PhD, Principal Investigator — University of Iowa
Locations (1):
- Institute for Health Reseach and Policy, UIC, Chicago, Illinois, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All recruitment took place online. A "No ad exposure" group was generated from program registrants, during a 4-week period (05/07/2012 - 06/03/2012) prior to the intervention.
  Recruitment for the "Ad exposure" intervention group took place during three 4-week periods: 06/04/2012 - 07/01/2012, 07/30/2012 - 08/26/2012, 09/24/2012 - 10/21/2012.
Groups:
- Ad Exposure: Young Adults, who register for the cessation program, by clicking through the online advertisements (intervention).
  Online advertisement : Internet advertisement with messages tailored for young adult smoker's motivated to quit
- No Ad Exposure: Young adults, who registered for the cessation program, after arriving at the program site though established means (e.g., search engine results), one month prior to presenting the tailored online advertisements (intervention).
Period: Overall Study
Arm/Group | Ad Exposure | No Ad Exposure
Started | 2676 | 394
Completed | 2676 | 394
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- No ad Exposure: Young adults, who registered for the cessation program, one month prior to presenting the online advertisements (intervention).
- Total: Total of all reporting groups
Arm/Group | Ad Exposure | No ad Exposure | Total
Number analyzed (Participants) | 2676 | 394 | 3070
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2676 | 394 | 3070
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | NA — This is a population internet-based study looking at overall cumulative rates of program enrollment; individual-level data were not collected. | NA — This is a population internet-based study looking at overall cumulative rates of program enrollment; individual-level data were not collected. | NA — Total not calculated because data are not available (NA) in one or more arms.
  Male | NA — This is a population internet-based study looking at overall cumulative rates of program enrollment; individual-level data were not collected. | NA — This is a population internet-based study looking at overall cumulative rates of program enrollment; individual-level data were not collected. | NA — Total not calculated because data are not available (NA) in one or more arms.
Region of Enrollment [Number; unit: participants]
  United States | 2676 | 394 | 3070

OUTCOME MEASURES:

1. Primary Outcome: Program Enrollment
Description: Rates of enrollment will be calculated as the proportion of visitors who enroll in treatment (e.g., number of enrollments/number of click-throughs from banner ads).
Time Frame: 1-month intervals over 7 months
Measure: Number; unit: proportion of click-throughs who enroll
Units Other Than Participants: Click-through from advertisements
Groups:
- Ad Exposure: Young Adults, who enrolled for the cessation program, by clicking through the online advertisements (intervention).
  Online advertisement : Internet advertisement with messages tailored for young adult smoker's motivated to quit
- No ad Exposure: Young adults, who enrolled for the cessation program, one month prior to presenting the online advertisements (intervention).
Arm/Group | Ad Exposure | No ad Exposure
Number analyzed (Participants) | 2676 | 394
Number analyzed (Click-through from advertisements) | 52260 | 0
proportion of click-throughs who enroll | .05 |

ADVERSE EVENTS:
Description: Serious and/or other [non-serious] events were not collected/assessed.
Arm/Group | Ad Exposure | No ad Exposure
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No